CLINICAL TRIAL: NCT01115582
Title: Open Label, Single Center, Nonrandomized Study Comparing Efficacy of To Be Marketed Cholic Acid With That of the Currently Used Formulation of Cholic Acid Capsules Used to Treat Children With Inborn Errors of Bile Acid Synthesis
Brief Title: Efficacy of To Be Marketed (TBM) Cholic Acid Capsules Used to Treat Children With Inborn Errors of Bile Acid Synthesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAC-001-01
Record Dates: First submitted 2010-01-19; First posted 2010-05-04 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Inborn Errors of Bile Acid Synthesis
Keywords: Inborn Errors; Bile Acid; Pediatrics; Liver Disease
MeSH Terms: conditions — Liver Diseases | interventions — Cholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholic Acid Capsule (Experimental): Manufactured cholic acid capsules
  Interventions: Drug: Cholic acid

INTERVENTIONS:
Drug: Cholic acid — The IUPAC name for cholic acid is 3 alpha,7alpha,12 alpha-trihydroxy-5 beta-cholanoic acid. The international nonproprietary name (INN) is cholic acid.
  Each patient will be given a box containing a 1 month supply of study drug. Each bottle will contain 90 capsules; each capsule will contain either 50 or 250 mg of manufactured cholic acid depending upon the child's weight. The study drug will be taken orally, in divided doses (as determined by the investigator), for a total daily dose of 10-15 mg/kg body weight. Parents of infants and young children who are unable to swallow the TBM cholic acid capsule will be instructed to sprinkle the contents of the capsule over 1-2 teaspoons of plain applesauce and feed it to the child.

SUMMARY:
This is a study in a small population of children who have inborn errors of bile acid synthesis who are currently taking established doses of the currently used cholic acid capsules prepared at the Cincinnati Children's Hospital Pharmacy. The study is designed to compare the efficacy of these currently used capsules with the efficacy of the same treatment provided in a cholic acid capsule that is made by a company that will be marketed after FDA approval.

At baseline, patients receive established doses of cholic acid capsules prepared at the Cincinnati Children's Hospital Medical Center Pharmacy. During the study, patients receive the same treatment provided in the to-be-marketed (TBM) cholic acid capsule. Hence, patients serve as their own controls, with baseline values presenting the reference value (CCHMC cholic acid capsule) and values after 30 days treatment presenting the value for the investigational treatment (TBM cholic acid capsule).

DETAILED DESCRIPTION:
Bile acids are end products of cholesterol metabolism. Individuals with inborn errors of bile acid synthesis lack the enzymes needed to synthesize the primary bile acids cholic acid and chenodeoxycholic acid (CDCA). These conditions are serious and account for approximately 1% of cases presenting as idiopathic cholestatic liver disease. The liver disease associated with these inborn errors in bile acid synthesis is progressive and, if untreated, may lead to death from cirrhosis and liver failure.

Monotherapy with cholic acid is considered the most appropriate therapeutic strategy to treat inborn errors in bile acid synthesis because it provides a stimulus for bile flow and inhibits endogenous production and accumulation of potentially hepatotoxic and cholestatic bile acid precursors, while additionally facilitating the absorption of fats and fat-soluble vitamins. At therapeutic doses, adverse effects are not generally observed and as such, cholic acid has become the treatment of choice at the Cincinnati Children's Hospital since 1994.

This study will bridge data on the effectiveness of a standardized manufactured preparation to data obtained from patients originally treated with the currently used cholic acid capsules formulated in the CCHMC Pharmacy before being switched to the manufactured preparation.

ELIGIBILITY:
Inclusion Criteria:

* must have stable transaminase levels within 2 times the upper limits of the normal range.
* must have a diagnosis of an inborn error of bile acid synthesis.
* must have signed the written informed consent/assent document before study start.
* must be currently receiving currently used cholic acid therapy under IND 45,470.
* must be willing and able to comply with all study assessments and procedures.
* must be able to make two visits (Visit 1 and Visit 2) to the study site.

Exclusion Criteria:

* is not currently receiving cholic acid therapy for inborn errors of bile acid synthesis under IND 45,470.
* is unable or unwilling to comply with study requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Heubi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Bove KE, Heubi JE, Balistreri WF, Setchell KD. Bile acid synthetic defects and liver disease: a comprehensive review. Pediatr Dev Pathol. 2004 Jul-Aug;7(4):315-34. doi: 10.1007/s10024-002-1201-8. Epub 2004 Jul 15. PMID 15383928
- [Background] Gonzales E, Gerhardt MF, Fabre M, Setchell KD, Davit-Spraul A, Vincent I, Heubi JE, Bernard O, Jacquemin E. Oral cholic acid for hereditary defects of primary bile acid synthesis: a safe and effective long-term therapy. Gastroenterology. 2009 Oct;137(4):1310-1320.e1-3. doi: 10.1053/j.gastro.2009.07.043. Epub 2009 Jul 19. PMID 19622360
- [Background] Heubi JE, Setchell KD, Bove KE. Inborn errors of bile acid metabolism. Semin Liver Dis. 2007 Aug;27(3):282-94. doi: 10.1055/s-2007-985073. PMID 17682975
- [Background] Jacquemin E., Gerhardt M, Cresteil D, Fabre M, Taburet AM, Hadchouel M, Trivin F, Stechell KDR and Bernard O. Long-term effects of bile acid therapy in children with defects of primary bile acid synthesis: 3ß-Hydroxy-C27-steroid dehydrogenase/isomerase and Delta4-3-Oxosteroid 5ß-reductase deficiencies. In: van Berge Henegouwen GP, et al. (eds): Falk Symposium No 120: Biology of Bile Acids in Health and Disease. Kluwer Academic Publishers, Dordrecht/Boston/London; 2001:278-282.
- [Background] Setchell KD, Heubi JE. Defects in bile acid biosynthesis--diagnosis and treatment. J Pediatr Gastroenterol Nutr. 2006 Jul;43 Suppl 1:S17-22. doi: 10.1097/01.mpg.0000226386.79483.7b. PMID 16819396
- [Background] Setchell KDR, et al. A unique case of cerebrotendinous xantomatosis presenting in infancy with cholestatic liver disease further highlights bile acid synthetic defects as an important category of metabolic liver disease. In: van Berge Henegouwen GP et al. (ed): Falk Symposium No. 120: Biology of Bile Acids in Health and Disease. Boston: Kluwer Academic Publishers; 2001.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this single-arm study, patients served as their own controls: Reference was presented by the baseline value, when patients received cholic acid capsules prepared by the Cincinnati Children's Hospital Medical Center; Investigational Treatment was the to-be-marketed (TBM) cholic acid capsule administered to patients for 30 days treatment duration.
Pre-assignment Details: The study was performed in patients with inborn defects of bile acid synthesis currently receiving cholic acid capsules prepared by the Cincinnati Children's Hospital Medical Center (CCHMC) under IND 45,470. The study planned to include 25 patients; but only 16 patients fulfilled eligibility criteria and were willing to travel to the CCHMC.
Groups:
- Cholic Acid: All patients entered and treated
Period: Overall Study
Arm/Group | Cholic Acid
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Serum Transaminases
Description: Concentration of serum alanine transaminase (ALT) and aspartate transaminase (AST)
Time Frame: At baseline and after 30 days of treatment
Population: All patients entered and treated
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
U/L
  ALT, baseline | 31.4 (21.9)
  ALT, Day 30 | 30.9 (24.0)
  AST, baseline | 62.7 (27.1)
  AST, Day 30 | 65.0 (39.0)

2. Primary Outcome: Serum and Urine Bile Acids
Description: Concentration of bile acids in serum (S) and urine (U). (abbreviations: chol.=cholenoic; monohydro=monohydroxy; dihydro=monohydro)
Time Frame: At baseline (BL) and after 30 days of treatment (D30)
Population: All patients entered and treated
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
mmol/L
  U, BL: 3β,7α-dihydroxy-Δ5 sulfate m/z 469 | 12.37 (35.31)
  U, D30: 3β,7α-dihydroxy-Δ5 sulfate m/z 469 | 2.762 (3.955)
  U, BL: 3β,7α,12α-trihydroxy-Δ5 sulfate m/z 485 | 14.11 (42.78)
  U, D30: 3β,7α,12α-trihydroxy-Δ5 sulfate m/z 485 | 2.011 (2.995)
  U, BL: 3β,7α-dihydroxy-Δ5 gluycosulfate m/z 526 | 159.85 (474.52)
  U, D30: 3β,7α-dihydroxy-Δ5 gluycosulfate m/z 526 | 19.958 (29.341)
  U,BL: 3β,7α,12α-trihydroxy-Δ5 glycosulfate m/z 542 | 105.43 (337.05)
  U,D30: 3β,7α,12α-trihydroxy-Δ5 glycosulfate m/z542 | 5.421 (7.633)
  S,BL: Glyco-3-oxo-7-α,12α-dihydroxy-4-chol. m/z460 | 0.15 (0.07)
  S,D30: Glyco-3-oxo-7-α,12α-dihydroxy-4-chol.m/z460 | 0.055 (0.078)
  S,BL:Glyco-3-oxo-7-α,12α-monohydroxy-4-chol.m/z444 | 0.14 (0.01)
  S,D30:Glyco-3-oxo-7-α,12α-monohydro.-4-chol.m/z444 | 0.140 (0.184)
  S, BL: Tauro-3-oxo-7-α,12α-dihydroxy-4-chol.m/z510 | 0.52 (0.23)
  S,D30: Tauro-3-oxo-7-α,12α-dihydroxy-4-chol.m/z510 | 0.490 (0.679)
  S,BL:Tauro-3-oxo-7-α,12α-monohydroxy-4-chol.m/z498 | 0.05 (0.04)
  S,D30:Tauro-3-oxo-7-α,12α-monohydro.-4-chol.m/z498 | 0.020 (0.028)
  U, BL: Total 3β-hydroxy-Δ5 bile acids | 291.77 (889.56)
  U, D30: Total 3β-hydroxy-Δ5 bile acids | 30.148 (43.582)
  S, BL: Total 3-oxo-Δ4 bile acids | 0.84 (0.13)
  S, D30: Total 3-oxo-Δ4 bile acids | 0.705 (0.601)

3. Secondary Outcome: Adverse Events
Description: Total number of patients with any adverse events
Time Frame: Total of 30 days, i.e. from the time point the patients entered into the study up to the end of treatment
Population: All patients entered and treated
Measure: Number; unit: participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
participants | 9

4. Secondary Outcome: Blood Pressure
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP)
Time Frame: At baseline and after 30 days of treatment
Population: All patients entered and treated
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
mmHg
  SBP, baseline | 106.9 (10.2)
  SBP, Day 30 | 109.6 (6.6)
  DBP, baseline | 63.9 (6.7)
  DBP, Day 30 | 65.4 (6.8)

5. Secondary Outcome: Physical Examination
Description: Total number of patients with abnormal findings from general physical examination
Time Frame: At baseline (BL) and after 30 days of treatment (D30)
Population: All patients entered and treated
Measure: Number; unit: participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
participants
  BL, N patients with abnormal physical findings | 0
  D30, N patients with abnormal physical findings | 0

6. Secondary Outcome: Total Bilirubin
Description: Concentration of total bilirubin in serum
Time Frame: At baseline and after 30 days of treatment
Population: All patients entered and treated
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cholic Acid
Number analyzed (Participants) | 16
mg/dL
  Baseline, total bilirubin | 0.35 (0.37)
  D30, total bilirubin | 0.32 (0.28)

ADVERSE EVENTS:
Time Frame: Total of 30 days, i.e. from the time point the patients entered into the study up to the end of treatment
Arm/Group | Cholic Acid
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cholic Acid (N=16)
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cholic Acid (N=16)
Decreased/low 250H/Vit D (General disorders) | 4
Decreased Vitamin A (General disorders) | 1
Nosebleed (Vascular disorders) | 1 — In the clinical study Report, the Event was counted towards the Body System "Eye, ear, nose, throat"
Diarrhoea (Gastrointestinal disorders) | 1
Reflux (Gastrointestinal disorders) | 1
Increased ALT (Hepatobiliary disorders) | 1
Increased AST (Hepatobiliary disorders) | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No